CLINICAL TRIAL: NCT00040430
Title: Study of 111In-DAC as a Medical Imaging Agent for the Detection of Breast Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Copharos (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CP101
Record Dates: First submitted 2002-06-26; First posted 2002-06-28 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

INTERVENTIONS:
Drug: 111In-DAC
Procedure: Diagnostic

SUMMARY:
The purpose of this study is to investigate the safety and imaging ability of 111In-DAC when used with planar and SPECT imaging for the detection of breast cancer.

ELIGIBILITY:
Inclusion Criteria

Patients will be eligible for the study if they:

* Are non-pregnant, non-lactating females 18 years of age or older(must agree to use an appropriate and effective method of birth control during the study and for 2 weeks after study)
* Are being evaluated for a known or suspected breast tumor (must present with either a mammographic abnormality 10mm or larger or a mammographically occult but palpable abnormality of the breast)
* Have been previously scheduled for biopsy or surgical excision of the known or suspected tumor of the breast
* Have signed an informed consent form

Exclusion Criteria

Patients will not be eligible for this study if they:

* Have a history or suspicion of significant allergic reaction or anaphylaxis to any of the 111In-DAC components
* Have a clinically unstable medical condition or opportunistic infection, a life-threatening disease state, impaired renal or hepatic function or are immunosuppressed
* Are taking or have taken part in any investigational study within 30 days of start of study
* Have received an indium agent within 30 days of start of study
* Are not able to remain immobile during scanning time
* Have taken drugs that may damage the kidneys within 2 weeks of start of study
* Have abnormal laboratory test results: hemoglobin < 9.5 gms/dl, serum creatinine > 1.5 mg/100ml, alkaline phosphatase 2X the upper limit of normal
* Have undergone an excisional and/or needle localization biopsy within 4 days prior to start of study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Sutter Roseville Medical Center, Roseville, California
  - University at Buffalo, Buffalo, New York